CLINICAL TRIAL: NCT04261517
Title: Efficacy and Safety of Hydroxychloroquine for Treatment of COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Hongzhou Lu, professor, Shanghai Public Health Clinical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HC-COVID-19
Record Dates: First submitted 2020-02-06; First posted 2020-02-07 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Pneumonia, Pneumocystis; Coronavirus; COVID-19
Keywords: Pneumonia; COVID-19; hydroxychloroquine
MeSH Terms: conditions — Pneumonia, Pneumocystis; Coronavirus Infections; COVID-19; Pneumonia | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine and conventional treatments (Experimental): After randomization, subjects take hydroxychloroquine 400mg per day for 5 days, also take conventional treatments.
  Interventions: Drug: Hydroxychloroquine
- Conventional treatments (No Intervention): After randomization, subjects take conventional treatments without hydroxychloroquine.

INTERVENTIONS:
Drug: Hydroxychloroquine — Subjects take hydroxychloroquine 400 mg per day for 5 days, also take conventional treatments
  Arms: Hydroxychloroquine and conventional treatments

SUMMARY:
The study aims to evaluate the efficacy and safety of hydroxychloroquine in the treatment of COVID-19 pneumonia.

DETAILED DESCRIPTION:
There is no vaccine or antiviral treatment for human coronavirus, so this study aims to evaluate the efficacy and safety of hydroxychloroquine in the treatment of COVID-19 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* The participants were diagnosed as COVID-19 pneumonia, according to the notice on printing and distributing the diagnosis and treatment plan of pneumonia with new coronavirus infection (trial version 4 or update version) made by National Health Commission of the People's Republic of China;
* Participants aged over 18;
* Written the informed consent.

Exclusion Criteria:

* Hypersensitivity to chloroquine or hydroxychloroquine;
* Women during pregnancy;
* Severe heart, lung, kidney, brain, blood diseases or other important systemic diseases;
* Participants with retinal disease, hearing loss;
* Participants with severe neurological and mental illness;
* Subjects were considered to be unable to complete the study, or not suitable for the study by researchers.

Exit criteria:

* Subjects asked to withdraw the study
* Subject will benefit if withdraw according to researchers' suggestions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
The virological clearance rate of throat swabs, sputum, or lower respiratory tract secretions at day 3 | 3 days after randomization
The virological clearance rate of throat swabs, sputum, or lower respiratory tract secretions at day 5 | 5 days after randomization
The virological clearance rate of throat swabs, sputum, or lower respiratory tract secretions at day 7 | 7 days after randomization
The mortality rate of subjects at weeks 2 | 14 days after randomization

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 14 days after randomization
The critical illness rate of subjects at weeks 2 | 14 days after randomization
  The diagnosis of critical illness case was based on the notice on printing and distributing the diagnosis and treatment plan of pneumonia with new coronavirus infection (trial version 4) made by National Health Commission of the People's Republic of China.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen J, Liu D, Liu L, Liu P, Xu Q, Xia L, Ling Y, Huang D, Song S, Zhang D, Qian Z, Li T, Shen Y, Lu H. [A pilot study of hydroxychloroquine in treatment of patients with moderate COVID-19]. Zhejiang Da Xue Xue Bao Yi Xue Ban. 2020 May 25;49(2):215-219. doi: 10.3785/j.issn.1008-9292.2020.03.03. Chinese. PMID 32391667
- See also: The results have been published on the Journal of Zhejiang University (Medical Sciences) — http://www.zjujournals.com/med/CN/10.3785/j.issn.1008-9292.2020.03.03